CLINICAL TRIAL: NCT02749734
Title: Clinical Study of Subretinal Transplantation of Human Embryo Stem Cell Derived Retinal Pigment Epitheliums in Treatment of Macular Degeneration Diseases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, ZhengQin Yin, Professor, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013CB967002
Record Dates: First submitted 2016-01-07; First posted 2016-04-25 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Macular Degeneration; Stargardt's Macular Dystrophy
Keywords: Human embryo stem cell derived retinal pigment epitheliums; Subretinal transplantation; Wet Age related Macular degeneration; Stargardt's macular dystrophy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hESC-RPE (Experimental): Subretinal transplantation of Human embryo stem cell derived retinal pigment epitheliums
  Interventions: Procedure: Subretinal transplantation

INTERVENTIONS:
Procedure: Subretinal transplantation — Transplant hESC-RPE into subretinal space of patients with macular degeneration

SUMMARY:
The purpose of this study was to determine the safety and therapeutic effect of sub-retinal transplantation of human embryo stem cell derived retinal pigment epitheliums (hESC-RPE) in patients with macular degeneration diseases, and explore new treatment modalities for macular degeneration diseases (Age-related macular degeneration and Stargardt's macular dystrophy).

ELIGIBILITY:
Inclusion Criteria:

* Aging from 18 to 75 years
* must have signed informed consent
* At least one visually impaired eye caused by macular degeneration diseases
* Can not be effectively treated with conventional therapies
* Best corrected visual acuity scores between 19 and 73 letter in ETDRs (early treatment diabetic retinopathy ) eye chart , including 19 and 73 (or the equivalent of Snellen eyesight from 20/400 to 20/40)
* Visual loss caused by macular degeneration diseases

Exclusion Criteria:

* Eyes with concomitant diseases which will interfere the visual improvement of the study
* Active intraocular inflammation regardless of the grade of severity
* Active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, ophthalmia)
* History of uveitis
* Severe cataract, glaucoma, retinal blood vessels occlusion, retinal detachment, macular hole, vitreous-macula traction
* Iris neovascularization
* Patients who have only one functioning eye, or the best corrected vision of untreated eye scores less than 24 letters in ETDRS chart(corresponding to 20/320 in Snellen chart)
* History of intraocular surgery
* Severe systemic diseases: Stroke, coronary heart disease, angina pectoris, renal insufficiency needing dialysis
* Allergic to sodium fluorescein
* Uncontrolled hypertension (systolic pressure>140mmHg,or diastolic pressure>90mmHg)
* Coagulative function disorder
* System administration of drugs that are toxic to lens, retina, or optic nerve like hydroxychloroquine, phenothiazine, ethambutol, tamoxifen, etc.
* Involved in other clinical trials of any medicine within 1 month (or within 5 half-life periods)
* Have maternity plan in 6 months
* In pregnancy or lactation period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-Related Adverse Events [Safety and Tolerability] | up to 12 months
  Patients with Treatment-Related Adverse Events caused by local rejection of implanted cells or systemic immunosuppression treatment

SECONDARY OUTCOMES:
Number of Early Treatment Diabetic Retinopathy (ETDR ) letters participants can recognize | up to 12 months
  Visual acuity is reflected by number of ETDR letters participants can recognize
Visual Field as examined by Static perimetry | up to 12 months
  Area and sensitivity of visual field are detected by Static perimetry
Flash Electroretinogram (FERG) | up to 12 months
  Retinal electrophysiological function is tested by FERG
Amplitude and Latency of Flash Visual Evoked Potentials (FVEP) | up to 12 months
  Optic nerve function as assessed by FVEP
Multifocal Electroretinogram (MFERG) | up to 12 months
  Local retinal function as assessed by MFERG

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Lv YX, Li QY, Duan P, Zhang MF, Liu B, Li SY, Zhao TT, Wang H, Liu Y, Yin ZQ. Safe CNV removal is crucial for successful hESC-RPE transplantation in wet age-related macular degeneration. Stem Cell Reports. 2025 Mar 11;20(3):102424. doi: 10.1016/j.stemcr.2025.102424. Epub 2025 Feb 27. PMID 40020685